CLINICAL TRIAL: NCT07042776
Title: Satisfaction and Feasibility Evaluation of an Electronic Massager (Expert Manipulative Massage Automation -EMMA) Compared to Massage Therapist-delivered Massage
Brief Title: Satisfaction and Feasibility Evaluation of an Electronic Massager Compared to Massage Therapist-delivered Massage
Acronym: EMMA2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 25-002916
Record Dates: First submitted 2025-06-05; First posted 2025-06-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Massage Therapy
Keywords: EMMA; Expert Manipulative Massage Automation; Massage Therapy; EMMA@TREATMENT

STUDY DESIGN:
Intervention Model Description: Two different massage therapies will be experienced by subjects: EMMA electronic massage and massage therapy by a massage therapist. The order in which the massages will be experienced will be determined by randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EMMA treatment, then therapist-delivered massage (Experimental): Subjects in this arm will first undergo massage therapy utilizing the EMMA Massager (Expert Manipulative Massage Automation). A minimum of 24 hours later, the subjects will undergo a massage therapist-delivered massage.
  Interventions: Device: EMMA (Expert Manipulative Massage Automation); Other: Therapist-delivered massage
- Therapist-delivered massage, then EMMA treatment (Experimental): Subjects in this arm will first undergo a massage therapist-delivered massage treatment. A minimum of 24 hours later, the subjects will undergo massage therapy utilizing the EMMA Massager (Expert Manipulative Massage Automation).
  Interventions: Device: EMMA (Expert Manipulative Massage Automation); Other: Therapist-delivered massage

INTERVENTIONS:
Device: EMMA (Expert Manipulative Massage Automation) — For the EMMA massage, the subject lies down on the robot platform in a prone position. A therapist sets the robot parameters. The EMMA electronic massager applies massage to the focus points on the back of the participants guided by cameras and computer programs. Treatment lasts approximately 20-30 minutes.
Other: Therapist-delivered massage — For the therapist-delivered massage treatment, the licensed massage therapist will follow standard of care protocol. Treatment lasts approximately 20-30 minutes.

SUMMARY:
The objective of this study is to evaluate the practicality and acceptability of using an electronic massager. Additionally, it aims to compare user satisfaction between the experience with an electric massager and a massage provided by a professional massage therapist.

DETAILED DESCRIPTION:
This study is being done to understand how practical and acceptable EMMA, an electronic massage device, is, and the satisfaction of the EMMA massage compared to massage therapy given by a certified massage therapist. Participants will also be asked to have two massages, one given by EMMA and another delivered by a massage therapist. The order in which participants will receive each massage will be determined by randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability to provide informed consent
* Women of childbearing potential who self-report not being pregnant and agree to employ an effective method of birth control (surgical sterilization or oral contraceptives, barrier method with spermicides, intrauterine device, etc.) during the study period
* Ability to complete all aspects of this trial

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients with inability of staying in a prone position
* Patients with bleeding disorders
* Patients with a current diagnosis of cancer or being treated for cancer
* Patients with allergies and/or local skin affectations
* An unstable medical or mental health condition as determined by the physician investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients enrolled | Duration of study, approximately 2 years
  Feasibility will be determined by the total number of patients screened in order to accrue the 40 needed to complete the study.

CONTACTS AND LOCATIONS:
Overall Officials: Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No